CLINICAL TRIAL: NCT02676453
Title: Dental Hygienist Support Promotes Good Oral Health in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Dental Health, Varmland (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VarmlandBL
Record Dates: First submitted 2016-02-01; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Impaired Health
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Dental hygienist support
  Interventions: Other: Intervention
- control (No Intervention): Care as usal

INTERVENTIONS:
Other: Intervention — Dental hygienist support
  Arms: Intervention

SUMMARY:
Objective: The aim of this study was to evaluate the effects of dental hygienist support on oral health and attitudes to oral healthcare in nursing homes for older people.

Background: Studies in long-term care facilities have indicated that oral health is often unsatisfactory. It is important that nursing staff are able to assist dependent care recipients. Dental hygienist support has been suggested as valuable help.

Material and methods: Two nursing homes were randomly selected for intervention and control. Interventions included weekly support from dental hygienists on oral hygiene procedures, prescriptions for individual oral hygiene procedures, and oral care organisational issues. The residents' oral health, measured by dental plaque levels, gingival bleeding and the Revised Oral Assessment Guide (ROAG), was evaluated before and after three months. Attitudes among the staff to oral healthcare were collected through a questionnaire.

DETAILED DESCRIPTION:
Introduction Oral health in older people has been the subject of several studies from different perspectives in recent decades. These studies describe the difficulties in achieving a holistic view in healthcare when it comes to oral health for older people, and a lack of awareness among nursing staff that infections in the oral cavity may also affect other parts of the body. In a randomised study, it was shown that professional oral healthcare may improve oral conditions in elderly people. Studies have shown correlations between poor oral hygiene and pneumonia in elderly people. It has also been shown that both chewing ability and daily nutritional intake may be adversely affected in individuals with partial or full dentures compared to those with natural teeth or crown and bridge work.

To ensure good oral health and function, it is of great importance that nursing staff are able to support dependent older people in their daily oral care. Basic oral health knowledge among nursing staff and further training in oral hygiene procedures have been reported to be essential to good quality in oral care. In a study from Norway, it was shown that the residents' oral hygiene in nursing homes was significantly improved when an oral healthcare program was introduced. The program consisted of new procedures and tools for good oral hygiene, as well as practical training in oral care for nursing staff.

An earlier study by the authors of the present study captured the views of staff in various nursing homes for older people on important aspects for well-functioning daily oral care for residents. This study emphasised organisational structures involving oral hygiene procedures, staff approach regarding prioritising oral hygiene and keeping up skills in oral hygiene procedures, and staff views on residents' needs including matters such as how to act when a resident refuses help with oral care. Support by a dental hygienist in the nursing home was perceived as valuable help. Other authors have made similar findings in long-term care facilities, indicating that oral hygiene may be unsatisfactory due to organisational factors such as lack of a standard protocol for oral hygiene procedures, lack of time and conflicting priorities, lack of knowledge among care providers and cooperation difficulties among some residents.

The aim of the present study was to evaluate the effects of dental hygienist support on oral health and attitudes to oral health care in nursing homes for older people.

Material and Methods The study had a quantitative design with two comparable study groups with older people in two nursing homes. The two most centrally situated public nursing homes in the largest municipality in the county of Värmland in Sweden were randomly selected as intervention and control group. The Regional Ethical Review Board in Uppsala approved the study.

Study material The two nursing homes were comparable regarding size, resident profile, and staffing. The residents included older people with dementia, physical disabilities or long-term illnesses. One director of nursing, one registered nurse and 21 nursing assistants worked at the intervention nursing home. One director of nursing, one registered nurse and 28 nursing assistants worked at the control nursing home. All but one of the staff members were women. There were 33 residents in each of the two nursing homes. Only dentate residents were included.

Procedures The Director of Social Services in the municipality was given verbal and written information and approved the study. The directors of nursing at the intervention and control nursing homes were separately informed, both verbally and in writing, about the procedures for their respective part of the study. They were not informed which additional nursing home was participating in the study. The directors of nursing at both nursing homes supplied the residents or their relatives with written information about the study and asked for written consent. Only those who consented to participate in the study were included. Edentulous residents were excluded from the study. The nursing assistants agreed to participate in the study.

Intervention

In the intervention nursing home, the study dental hygienists offered regular support over the course of three months, comprising the following:

* Participation in staff meetings with the director of nursing and nursing assistants at the beginning of the study, after six weeks and at the end of the study period. At those meetings, oral care routines were discussed and a concept of prescriptions for individual oral hygiene procedures was introduced (see below).
* Visits to the nursing home once a week. For two hours in the morning, the dental hygienists accompanied and supported the nursing staff in their oral hygiene care and gave advice on daily oral hygiene procedures for each resident participating in the study. Specific difficulties concerning residents with cooperation problems were addressed. Each weekly visit ended with a 30 min meeting in which the nursing staff had the opportunity to discuss oral hygiene procedures and oral health issues with the dental hygienists.
* Individual written oral hygiene prescriptions for special oral hygiene devices, procedures or products. These were issued by the dental hygienists to residents with an identified need for extra oral care support, i.e. with scores >1 in the Revised Oral Assessment Guide (ROAG) evaluation.

Control

At study start, the director of nursing for the control nursing home was informed about the importance of good oral hygiene and was invited to contact the two study dental hygienists if support was needed with any particular oral health issue or dental hygiene procedure.

Clinical evaluation of oral health Clinical evaluations of the residents' oral health status were blinded. An independent dentist and dental hygienist, otherwise not committed to the planning of the study and not informed about which was the intervention nursing home, conducted a dental examination of the residents who had consented to take part in the study in both nursing homes. This was done at the beginning of the study and three months later at the end of the study. The staff were not informed about the scheduled time for the clinical evaluations of the residents' oral health.

ELIGIBILITY:
Inclusion Criteria:

* Residents at a nursing home
* Natural teeth

Exclusion Criteria:

* Edentulous

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in dental plaque levels after three months | 3 months
  Four surfaces (proximal, buccal and lingual surfaces) on each tooth is measured and regarding dental plaque in four levels.
Changes in gingival bleeding levels after three months | 3 months
  Four surfaces (proximal, buccal and lingual surfaces) on each tooth is measured and regarding gingival bleeding in four levels.

SECONDARY OUTCOMES:
Changes in Revised Oral Assessment Guide, ROAG, after 3 months | 3 months
  ROAG includes assessment of voice, lips, oral mucosa, tongue, gums, teeth, dentures, saliva and swallowing ability. Each item was rated according to a ROAG score of 1 (normal), 2 (minor problems) and 3 (severe problems). Definitions are given for each item in ROAG. For example, the item "teeth" includes the following definitions: 1 (normal) clean teeth, no visible plaque or food debris, 2 (minor problems) plaque or food debris in localised areas, 3 (severe problems) generalised plaque, food debris or defective teeth. The item "gums" includes the following definitions: 1 (normal) pink and firm, 2 (minor problems) edematous with or without redness, 3 (severe problems) spontaneous bleeding. The item "lips" includes: 1 (normal) smooth, pink, moist, 2 (minor problems) dry or cracked, angular cheilitis, 3 (severe problems) ulcerated or bleeding.

OTHER OUTCOMES:
Intervention staff evaluation of oral health care at baseline assessed with a questionnaire | Only once at baseline
  Intervention nursing home staff was asked to fill in a questionnaire A. The questionnaire covered background information and questions including items on organisation and what to do when residents didn't cooperate graded on Likert-type four- or five-point scales.
Intervention staff evaluation of oral health care after 3 months assessed with a questionnaire | 3 months
  After three months, the nursing staff was asked to answer a modified version of questionnaire A, questionnaire B. Ten additional questions covered how the nursing staff had experienced their participation in the study. They evaluated if documentation and communication on oral care between staff members had improved and if their knowledge about and confidence in oral health care had been affected, all graded on a Likert-type four-point scale from "very little" to "yes, absolutely".

CONTACTS AND LOCATIONS:
Overall Officials: Inger Wårdh, DdS, PhD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No